CLINICAL TRIAL: NCT06606678
Title: The Role of Regular Physical Activity in Promoting Metabolic Health, Reducing Inflammation, and Improving Gut Function in Individuals Aged 50 Years and Older
Brief Title: The Role of Regular Physical Activity in Enhancing Metabolic Health, Reducing Inflammation, and Improving Gut Function
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 423/24
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Intestinal Inflammation; Metabolic Disease
Keywords: physical activity; metabolic health; inflammation; gut function; older adults
MeSH Terms: conditions — Metabolic Diseases; Motor Activity; Inflammation | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- excercise (Experimental): supervised excercise training; twice a week for 12 months
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — supervised exercise training; twice a week for 12 months

SUMMARY:
The goal of this clinical trial is to learn if regular physical activity can improve metabolic health, reduce inflammation, and decrease gut permeability in individuals aged 50 and older. The main questions it aims to answer are:

Does regular physical activity, even at low intensity, improve metabolic parameters? Does physical activity reduce inflammation and gut permeability in older adults? Researchers will compare a group participating in low-intensity dance classes to a group participating in higher-intensity calisthenics training to see if the intensity of exercise has different effects on these outcomes.

Participants will be asked to:

Attend organized training sessions led by instructors twice a week for 12 months.

Complete anthropometric measurements (height, weight) and body composition analysis (DXA scan).

Provide blood samples for biochemical analysis (glucose, insulin, CRP, etc.). Submit stool samples for gut health markers (calprotectin, zonulin, etc.). Complete surveys on lifestyle and dietary habits before and after the study.

DETAILED DESCRIPTION:
The project aims to assess the impact of increased physical activity on inflammation and gut permeability, and consequently on metabolic health in individuals.

Hypothesis: Regular physical activity, even at low intensity, improves metabolic parameters and reduces gut inflammation, thus positively affecting the health of individuals.

Description: The study will involve individuals aged 50 and older. The experimental group will consist of 50 participants who will engage in organized exercise sessions led by trainers twice a week for 12 months, and 50 participants who will not participate in sports activities. Participants will be assessed twice, before the start of the exercise program and after completing the 12 month training program. Participants will be recruited into two groups differing in training intensity. One group will participate in low-intensity dance classes, while the other group will engage in calisthenics (body weight resistance training) at a higher intensity.

The study will include: anthropometric measurements, body composition analysis, surveys, biochemical tests, and stool sample analysis. Height will be measured using a GMP Swiss Made anthropometer (accuracy ±1mm), body weight with an electronic personal scale RADWAG C315.60/150.OW-1 (accuracy ±100g), and body composition will be assessed using dual-energy X-ray absorptiometry (DXA) with the Lunar Prodigy device (General Electric Medical Systems, USA). Lifestyle and dietary habits will be assessed using a questionnaire method. The food frequency questionnaire (FFQ) and food diaries (participants will be asked to record their intake for 3 days before the start and 3 days after the completion of the training program) will be used.

Biochemical blood tests will measure glucose, insulin, amylin, C-peptide, ghrelin, glucose-dependent insulinotropic peptide (GIP), glucagon-like peptide-1 (GLP-1), leptin, and secretin as markers of metabolic changes, as well as C-reactive protein (CRP), calprotectin, zonulin, and secretory immunoglobulin A as markers of inflammation and gut permeability. The measurement of metabolic markers will be performed using commercially available Multiplex kits (based on magnetic bead technology), allowing for a broader range of results with a smaller volume of biological material and lower overall cost. The assessment of inflammation and gut permeability markers will be performed using commercially available ELISA kits. Based on fasting glucose and insulin levels, the insulin sensitivity index HOMA-IR will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Age over 50 years
* No contraindications for engaging in physical activity

Exclusion Criteria:

* Presence of diseases that prevent participation in physical activity

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in insulin sensitivity | before and after 12 months of intervention
  To assess the primary outcome measure of improvement in insulin sensitivity, we will use the HOMA-IR index.

SECONDARY OUTCOMES:
Reduction in gut inflammation | before and after 12 months of intervention
  Reduction in gut inflammation will be assessed by measuring decreases in biomarkers such as calprotectin, zonulin, and secretory immunoglobulin A in stool samples/blood samples using ELISA kits.

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Bryl, PhD, Study Director — Poznan Univeristy of Physical Education
Locations (1):
- Poznań University of Physical Education, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No